CLINICAL TRIAL: NCT01994135
Title: Effects of Carbohydrase-inhibiting Polyphenols on Glycaemic Response in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Hilda Nyambe, PhD candidate, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MEEC 12-037
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Hyperglycaemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reference food (Active Comparator): The reference food is white bread
  Interventions: Other: Reference food
- Test food dose 1 (Experimental): Test food dose 1 response will be compared to reference test food
  Interventions: Other: Test food dose 1
- Test food dose 2 (Experimental): Test food dose 2 response will be compared to reference test food as well as to test food dose 1
  Interventions: Other: Test food dose 2

INTERVENTIONS:
Other: Reference food — Reference food will be used to which test food samples will be compared to.
  Arms: Reference food
Other: Test food dose 1 — Will contain low dose of a mixture of polyphenols in addition to the reference food
  Arms: Test food dose 1
Other: Test food dose 2 — Will contain high dose (twice of the low dose) of a mixture of polyphenols in addition to the reference food
  Arms: Test food dose 2

SUMMARY:
Consumption of carbohydrate containing foods or sugary drinks brings about changes to the blood glucose levels. After a meal or drink, blood glucose levels rise until it reaches a peak concentration usually after 30 minutes. When the body senses the increase in blood glucose, a hormonal process involving insulin takes place to ensure that the glucose is taken up from the blood for storage and where it is needed for energy in the body. This process then brings about a decrease in the concentration of glucose until it reaches approximately the starting concentration. The original concentration of glucose is attained approximately 2 hours after eating or drinking a carbohydrate food or sugary drink respectively.

Different carbohydrates and sugary drinks have different effects on blood glucose response depending on the amount as well as the type of carbohydrate. Those that give rise to a high glucose response compared to a reference carbohydrate (usually glucose) are said to be high glycaemic index (GI) foods and those with a lower glucose response compared to a reference carbohydrate (usually glucose) are said to be low glycaemic index (GI) foods.(1)

Research has shown that diets that give rise to a high glucose response are associated with a number of abnormalities like increased metabolic syndrome (2). Metabolic syndrome mostly comprises of insulin resistance and glucose intolerance which gives an increased risk of type 2 diabetes. (3) It also gives rise to other conditions like high blood pressure (arterial hypertension), elevated blood insulin levels (hyper-insulinemia), elevated amounts of fat in the liver (fatty hepatosis) and elevated amounts of lipids in the blood (dyslipidemia). After type 2 diabetes become clinically apparent, the risk of cardiovascular disease also rises. (4) Research has also shown that foods/drinks which raise blood glucose levels gradually (low GI) rather than rapidly (high GI) have health benefits which include reducing the risk of metabolic syndrome (5). In vitro studies have shown that polyphenols found in fruits, vegetables and plant based foods have a positive effect on carbohydrate metabolism and can lower the blood glucose levels. (6)

This research will determine whether the presence of polyphenols in the diet has any lowering effect on the blood glucose levels and hence the glycaemic index of foods. This will be determined by asking volunteers to consume polyphenol rich drink/food together with white bread and determine the glycaemic response. The GI of bread will be determined initially as a reference.

Analysis will be done by measuring blood glucose response to white bread alone as reference and then to white bread with test sample containing polyphenols and then determine GI and see how the GI of bread will be affected. Other analyses to be done are plasma insulin, glucagon, gastric inhibitory polypeptide (GIP) and glucagon like peptides-1 (GLP-1) as they all relate to glycaemic response.

Study hypothesis is that glucose metabolism will be affected.

NOTE:

1. Only healthy participants undertook the study (Hence metabolic syndrome participants not part of the study)
2. Only glucose and insulin were analysed in the plasma (hence GIP, GLP-1 and glucagon not part of end points)

DETAILED DESCRIPTION:
The world health organisation has reported that over 220 million people suffer from diabetes worldwide and that by the year 2030, this number will be doubled. The WHO also reports that in 2004, about 3.4 million people died from high blood sugar (WHO fact sheet number 312, January 2011). About 90% of all diabetes cases is due to type II diabetes. Type 2 diabetes is largely due to overweight and lack of physical activity characterised by high glucose levels (hyperglycaemia).

In the human diet, the source of blood glucose are carbohydrates. Dietary carbohydrate is important to maintain glycaemic homeostasis and provides the most of the energy in the diets of most people. The control of blood glucose is a hormonal process and it is very important to human physiology. Hormonal processes involve the release of insulin from the β- cells of the pancreatic cells which stimulates the uptake of glucose after a meal, to other tissues either for utilisation (glycolysis) or to be stored in the liver as glycogen (glycogenesis). When blood glucose falls below normal, glucagon is secreted from the pancreatic α-cells and it promotes liver glucose production by inducing the generation of glucose from non carbohydrate substrates such as amino and fatty acids (gluconeogenesis) and the generation of glucose from glycogen (glycogenolysis). In addition to insulin and glucagon, there are gut hormones which also play a role in controlling plasma glucose concentrations in the body. The two important peptide hormones are called Glucagon like peptides-1 (GLP-1) and Gastric Inhibitory Polypeptide (GIP). They are said to have incretin activity (promotion of glucose dependent insulin secretion). GIP is secreted from the upper small intestines by the K cells and its primary function is to stimulate glucose-dependent insulin secretion by acting on pancreatic islets. It also stimulates glucagon and it is said to respond to the presence of nutrients (Seino et al., 2010). GLP-1 is secreted from the lower intestine and colon by the L cells following exposure to ingested nutrients. It also stimulates insulin secretion and biosynthesis but inhibits glucagon. GLP-1 is said to have other health and disease related functions (Marathe et al., 2013).

When the glucose homeostasis hormonal control fails, it entails high blood glucose levels (postprandial hyperglycaemia) which can lead to metabolic syndrome which includes obesity, impaired glucose tolerance (IGT), hypertension and dyslipidemia. Disturbance of glucose homeostasis can also lead to other symptoms such as inflammation and oxidative stress at the whole body level as well as disturbances of the functionality in several organs as well as diabetes (Hanhineva et al). Therefore, as much as carbohydrates are required in the human body as a major source of energy, too much in the diet can have adverse health effects especially the one with high glycaemic effect.

The proposed mechanism adapted from (Aston, 2006) of how carbohydrates may affect human health is that when there is a continual presence of high glycaemic index foods in the diet, this gives rise to postprandial glucose rise as well as high insulin demand to act on the high blood glucose levels in the blood. This is by the action of the hormones GIP and GLP-1 which stimulates insulin release when they sense the presence of nutrients. Postprandial glucose rise and high insulin demand may lead to insulin resistance which is the major component of metabolic syndrome. High insulin demand may also lead to β-cell failure which may also result in hyperglycaemia which is also a cause of insulin resistance. Insulin resitance and hyperglycaemia are risk factors for metabolic syndrome and diabetes type 2.

Scientific evidence suggest that postprandial hyperglycaemia in humans has a major role to play in health priorities like type 2 diabetes and blood glucose control. It has been reported that about 90% of all diabetes cases consist of type 2 diabetes. Apart from type I and type 2 diabetes, there are other related conditions which include pre-diabetes (impaired glucose tolerance (IGT) and impaired fasting glucose (IFG) as well as metabolic syndrome (obesity, hypertension and insulin resistance). It has been reported that pre-diabetes and metabolic syndrome increases the risk of developing cardiovascular disease and diabetes mellitus (Coutinho et al., 1999). The glycaemic index was originally proposed with the aim of managing diabetes. However, recent studies have shown that the GI has potential in the prevention of type 2 diabetes as well as in the treatment of metabolic syndrome. Research has shown that high GI diets are associated with increased risk of developing type 2 diabetes (Hodge et al., 2004) and (Steven et al., 2002). More research by (Mckeown et al., 2004) and (Scaglioni et al., 2004) have shown that high GI diet is associated with a number of abnormalities like increased metabolic syndrome and insulin resistance. In the same way, a low GI diet is said to improve insulin sensitivity but more research is needed to support this. A few studies like that of (Frost et al., 1996) have shown this to be the case. However it was observed that it was difficult to know whether this was as a result of improved insulin sensitivity, or improved insulin secretion or due to reduced rate of glucose absorption.

Having anything in the diet that can either slow down the digestion and absorption of carbohydrates can help reduce the risk (Barclay et al., 2008). Among others, two potential solutions are that of consumption of low glycaemic index foods or having ingredients in the diet that can reduce the glycaemic index of foods as well as postprandial blood glucose levels. The presence of inhibiting components in the diet that can reduce postprandial glucose can also be a solution to reducing the risk. Drugs like carbose are currently used in some countries for the management of type 2 diabetes which act by inhibiting carbohydrate digestive enzymes. However, the use of acarbose has side effects such as nausea, flatulence and diarrhoea. It has been reported that polyphenols also have the potential to inhibit the rise in blood glucose by hindering the rapid absorption of glucose (Hanhineva et al., Williamson, 2013).

A review by (Hanhineva et al.) reported that research using animal models as well as a limited number of human studies, have shown that polyphenols and polyphenol rich foods or beverages have the potential to affect postprandial glycaemic responses and fasting glycaemia as well as an improvement of acute insulin secretion and sensitivity. Other possible mechanisms as reported in the review by (Hanhineva et al.), include pancreatic β- cells stimulation to secrete insulin as well as activation of insulin receptors, modulation of the release of glucose from the liver as well as of intracellular signalling pathways and gene expression.

A recent review by (Williamson, 2013) concluded that it is very possible that the effects of polyphenols in the diet will affect glycaemic index of foods as well as postprandial glucose responses in humans. The two mechanisms highlighted by which this can be achieved being the inhibition of sugar metabolising enzymes as well as transporters. This potential action of polyphenols can thus be compared to that of acarbose which acts by the same mechanism and research in chronic intervention studies has shown that it reduces diabetes risk (Chiasson J. et al., 2002). The review by Williamson, 2013 also mentioned the possibility of different mechanisms being inhibited at the same time would give the most promising effects. Therefore, the most effect would be observed when more than one of the suggested pathways was inhibited.

This research has utilised available information from literature on in vitro studies carried out and we came up with a food polyphenol rich mixture (PRM) containing polyphenols that showed the highest inhibition towards carbohydrates digestion and absorption at different stages. The polyphenol rich breakfast food to be used as the test food will comprise of Green tea and a combination of four fruit extracts. For the test, the PRM is consumed together with bread containing 50g available carbohydrates and the control meal is composed of bread, sugars (fructose, sucrose and glucose) present in the fruit extracts with water. The polyphenol rich mixture constituents have been analysed in our laboratory for total polyphenol contents, specific polyphenols and for inhibitory potential to make sure that the test sample has the capacity to inhibit in vitro before they can be used in humans. The results obtained are good and justifies their use in the human study.

The study was approved by the University of Leeds Mathermatical and Physical Sciences (MAPs) ethical commitee with application number MEEC12-037. A total of 16 volunteers will need to complete the study and should be healthy and their fasting blood glucose levels fall within the healthy range of 4.3-5.9mmol/L.

The volunteers are scheduled to attend 4 visits, once per week for 4 weeks. During each of the four visits, the volunteer comes fasted in the morning and the fasting blood glucose is collected by a trained nurse. The volunteer is then given a test meal and blood samples are collected at 15, 30, 45, 60, 90, 120,150 and 180 minutes after the first bite of the test meal. On the first and last visit, they are saved with the reference meal which is composed of bread, water and sugars to compensate those found in the fruit extracts. On the third and fourth days, they consume test meals of either the low dose or high dose of green tea and fruit extracts in addition to bread. The blood samples are processed accordingly to obtain plasma and stored in the -80°C. Plasma samples will be analysed for concentrations of glucose, insulin, glucagon, GIP and GLP-1. The results will be used to plot the area under the curve and results obtained after consuming test meals will be compared to those obtained after consumption of control meals.

NOTE:

1. Only healthy participants undertook the study (Hence metabolic syndrome participants not part of the study)
2. Only glucose and insulin were analysed in the plasma (hence GIP, GLP-1 and glucagon not part of end points)

ELIGIBILITY:
Inclusion Criteria:

* Group 1 - Healthy subjects

Not diabetic Fasting glucose (blood glucose level before breakfast) 3.9 -5.9mmol/L Not on long term prescribed medication (except contraceptives) Not pregnant or lactating Not on special diet (for losing weight or fruit extracts supplements) Aged 18-75

Group 2 - Metabolic syndrome risk group

Not diabetic With fasting glucose (blood glucose level before breakfast) in the range of 6.0 - 8.0mmol/l Not on long term prescribed medication (except contraceptives) Not pregnant or lactating Not on special diet (for losing weight or fruit extracts) Aged 18-75

Exclusion Criteria:

* Group 1 - Healthy subjects

Not healthy Diabetic Fasting glucose (blood glucose level before breakfast) 3.9 -5.9mmol/L On long term prescribed medication (except contraceptives) Pregnant or lactating On special diet (for losing weight or fruit extracts supplements) Aged below 18years or above 75years

Group 2 - Metabolic syndrome risk group

Not diabetic With fasting glucose (blood glucose level before breakfast) above 8.0mmol/l On long term prescribed medication (except contraceptives) Pregnant or lactating On special diet (for losing weight or fruit extracts) Aged below 18years or above 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in Incremental Area Under the Curve for glucose and insulin | Blood will be collected at different time points within 3 hours, twice a week, for two weeks per volunteer

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, Study Chair — University of Leeds; Hilda Nyambe, Principal Investigator — University of Leeds
Locations (1):
- School of Food Science and Nutrition, Leeds, West Yorkshire, United Kingdom